CLINICAL TRIAL: NCT02975115
Title: The Catholic University of Korea Cancer Research Institute
Brief Title: Evaluating True PCR-negative Rate of Frontline Dasatinib in Early Chronic Phase CML for Therapeutic Harmonization
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Seoul St. Mary's Hospital (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Dong-Wook Kim, Director, Seoul St. Mary's Hospital
Other Study IDs: PCR-DEPTH
Record Dates: First submitted 2016-11-14; First posted 2016-11-29 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Chronic Myelocytic Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples Without DNA — Rest of RNA samples after Q-RT-PCR analysis
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: RQ-PCR RNA Analysis — Conventional Q-RT-PCR every 3 months

SUMMARY:
This study is designed to confirm the efficacy of dasatinib 100mg once daily in producing a complete molecular response and to prove a possibility of "Operational Cure" in CMR patients.

DETAILED DESCRIPTION:
This study also examines kinetics of complete molecular responses using new highly sensitive PCR based technology, digital PCR, which is reported to have a sensitivity down to 6 log reduction.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have Ph+ CML in CP
* newly diagnosed chronic phase CML, except hydroxyurea, anagrelide and within 7 days imatinib treatment
* Subjects must be enrolled in this study within approximately 3 months (90 days) after the date of first being diagnosed with CML. Subjects are allowed to have clonal chromosomal abnormalities in addition to the Philadelphia chromosome and remain eligible
* 0-2 ECOG Performance Status (PS) Score
* Adequate hepatic function test
* Adequate renal function test
* Adequate other organ functions
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy
* WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to the start of investigational product.
* Subjects agree to sign informed consent

Exclusion Criteria:

* WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least one month (4 weeks) before and for at least 1 month (4 weeks) after the last dose of study medication.
* WOCBP using a prohibited contraceptive method (Not applicable for this study).
* Women who are pregnant or breastfeeding.
* Women with a positive pregnancy test at enrollment or prior to administration of study medication.
* Men whose sexual partners are WOCBP, who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least one month (4 weeks) after completion of study medication.
* A serious uncontrolled medical disorder or active infection that would impair the ability of the subject to receive protocol therapy.
* Known pleural effusion at baseline.
* Uncontrolled or significant cardiovascular disease
* History of significant bleeding disorder unrelated to CML
* Prior chemotherapy for peripheral stem cell mobilization. (Prior collection of un-mobilized peripheral blood stem cells is permitted).
* Prior or concurrent malignancy
* Evidence of digestive dysfunction that would prevent administration of study therapy by mouth
* Uncontrolled diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed, CP-CML patients ≥ 18 years of age. Use of dasatinib for less than three weeks prior to study entry is allowed.
  Adult patients with a molecularly confirmed diagnosis of BCR-ABL positive CML in new CP who have not been treated with any myeloablative or interferon alpha therapy.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2013-11; Primary Completion 2016-11 (Actual); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Rate of CMR(complete molecular response) | 36 month
  Level of Bcr-Abl transcript (Conventional Q-RT-PCR)

SECONDARY OUTCOMES:
Rate of MMR(major molecular response) | 3,6,12,24 and 36 months
  Level of Bcr-Abl transcript (Conventional Q-RT-PCR)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Goh HG, Lin M, Fukushima T, Saglio G, Kim D, Choi SY, Kim SH, Lee J, Lee YS, Oh SM, Kim DW. Sensitive quantitation of minimal residual disease in chronic myeloid leukemia using nanofluidic digital polymerase chain reaction assay. Leuk Lymphoma. 2011 May;52(5):896-904. doi: 10.3109/10428194.2011.555569. Epub 2011 Feb 21. PMID 21338281